CLINICAL TRIAL: NCT05189314
Title: Clinical Outcomes and Quality of Life Measures After Surgical Resection and Radiofrequency Ablation of Benign Thyroid Nodules
Brief Title: RFA of Benign Thyroid Nodules: Clinical Outcomes and Quality of Life Study
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jennifer Kuo, Associate Professor, Columbia University
Other Study IDs: AAAS2141
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Nodules
Keywords: Radiofrequency Ablation
MeSH Terms: conditions — Thyroid Nodule | interventions — Thyroidectomy; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Thyroidectomy: Patients with benign thyroid nodules who undergo surgical resection
  Interventions: Procedure: Thyroidectomy
- RFA: Patients with benign thyroid nodules who undergo radiofrequency ablation
  Interventions: Device: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Thyroidectomy — Surgical Resection of thyroid nodules
  Groups: Thyroidectomy
Device: Radiofrequency Ablation — Radiofrequency Ablation of thyroid nodules
  Groups: RFA

SUMMARY:
The purpose of this observational research is to evaluate and compare clinical outcomes after treatment for symptomatic benign multinodular goiter (MNG) patients. This is a data collection study in which we ask participants to give access to information generated before and after treatment of their condition.

DETAILED DESCRIPTION:
Benign multinodular goiter (MNG) refers to an enlarged thyroid gland with nodules within it, frequently owing to iodine deficiency. It is the most common endocrine disorder worldwide.

Significant growths of nodules can cause symptomatic compressive symptoms such as dysphagia, dyspnea, or vascular compression of the neck vessels. On occasion, these nodules can develop autonomy and secrete excess thyroid hormone (toxic multinodular goiter). Surgical resection has been the preferred treatment option for symptomatic multinodular goiters and addresses both compressive symptoms as well as hyperthyroidism, but is associated with small, but not negligible risk of nerve injury, hypoparathyroidism, and may confer a risk of hypothyroidism and dependence on thyroid hormone supplementation.

Thermoablative methods that induce local thermodestruction leading to nodule shrinkage and improvement in local symptoms and hyperthyroidism have recently emerged as a possible alternative treatment approach for MNG. Monopolar radiofrequency ablation (RFA) is presently the best documented thermoablative technique. Although RFA of thyroid nodules specifically, is still considered investigational in the United States, RFA of thyroid nodules has been used by several centers globally (mainly in South Korea, Italy, China, and Austria) since 2006 with excellent clinical outcomes. In addition, RFA of other solid tumors is a commonly performed procedure in the United states and all RFA devices, including the device that we will use for the clinical care of these patients, are cleared by the FDA (New devices/technology to the market are approved, but devices that have a predicate device/technology that are already on the market only need to be cleared). In response to its increasing popularity, the Korean Society of Thyroid Radiology commissioned a Task Force to develop recommendations for the optimal use of radiofrequency ablation for thyroid tumors in 2012, and these recommendations were recently revised in 2017 and the American Association of Clinical Endocrinologists recently recommended that ultrasound guided thermal ablation treatments be considered for solid or mixed symptomatic benign thyroid nodules.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/=18 years old with benign thyroid nodules

Exclusion Criteria:

* cardiac arrhythmia
* pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients (>/=18 years) with benign, non-functional benign thyroid nodules
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Percent Volume Change of Nodules | 6 months and 12 months
  Percent Volume Change of Nodules: ((Volume (baseline) - Volume (*m*))/Volume(baseline))*100
Change in Thyroid Stimulating Hormone (TSH) | 6 months and 12 months
  Change in serum TSH
ThyPRO 39 Survey Score | 12 months
  The Thypro 39 is a survey assessing quality of life in patients with thyroid disease. Scores range from 0-100 with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Kuo, MD MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durante C, Costante G, Lucisano G, Bruno R, Meringolo D, Paciaroni A, Puxeddu E, Torlontano M, Tumino S, Attard M, Lamartina L, Nicolucci A, Filetti S. The natural history of benign thyroid nodules. JAMA. 2015 Mar 3;313(9):926-35. doi: 10.1001/jama.2015.0956. PMID 25734734
- [Background] de Rienzo-Madero B, Sabra JP, Gand E, Donatini G, Kraimps JL. Unilateral benign multinodular versus solitary goiter: Long-term contralateral reoperation rates after lobectomy. Surgery. 2019 Jan;165(1):75-79. doi: 10.1016/j.surg.2018.04.074. Epub 2018 Nov 8. PMID 30415868
- [Background] Kim YS, Rhim H, Tae K, Park DW, Kim ST. Radiofrequency ablation of benign cold thyroid nodules: initial clinical experience. Thyroid. 2006 Apr;16(4):361-7. doi: 10.1089/thy.2006.16.361. PMID 16646682
- [Background] Na DG, Lee JH, Jung SL, Kim JH, Sung JY, Shin JH, Kim EK, Lee JH, Kim DW, Park JS, Kim KS, Baek SM, Lee Y, Chong S, Sim JS, Huh JY, Bae JI, Kim KT, Han SY, Bae MY, Kim YS, Baek JH; Korean Society of Thyroid Radiology (KSThR); Korean Society of Radiology. Radiofrequency ablation of benign thyroid nodules and recurrent thyroid cancers: consensus statement and recommendations. Korean J Radiol. 2012 Mar-Apr;13(2):117-25. doi: 10.3348/kjr.2012.13.2.117. Epub 2012 Mar 7. PMID 22438678
- [Background] Kim JH, Baek JH, Lim HK, Ahn HS, Baek SM, Choi YJ, Choi YJ, Chung SR, Ha EJ, Hahn SY, Jung SL, Kim DS, Kim SJ, Kim YK, Lee CY, Lee JH, Lee KH, Lee YH, Park JS, Park H, Shin JH, Suh CH, Sung JY, Sim JS, Youn I, Choi M, Na DG; Guideline Committee for the Korean Society of Thyroid Radiology (KSThR) and Korean Society of Radiology. 2017 Thyroid Radiofrequency Ablation Guideline: Korean Society of Thyroid Radiology. Korean J Radiol. 2018 Jul-Aug;19(4):632-655. doi: 10.3348/kjr.2018.19.4.632. Epub 2018 Jun 14. PMID 29962870
- [Background] Gharib H, Papini E, Garber JR, Duick DS, Harrell RM, Hegedus L, Paschke R, Valcavi R, Vitti P; AACE/ACE/AME Task Force on Thyroid Nodules. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS, AMERICAN COLLEGE OF ENDOCRINOLOGY, AND ASSOCIAZIONE MEDICI ENDOCRINOLOGI MEDICAL GUIDELINES FOR CLINICAL PRACTICE FOR THE DIAGNOSIS AND MANAGEMENT OF THYROID NODULES--2016 UPDATE. Endocr Pract. 2016 May;22(5):622-39. doi: 10.4158/EP161208.GL. PMID 27167915
- [Background] Jeong WK, Baek JH, Rhim H, Kim YS, Kwak MS, Jeong HJ, Lee D. Radiofrequency ablation of benign thyroid nodules: safety and imaging follow-up in 236 patients. Eur Radiol. 2008 Jun;18(6):1244-50. doi: 10.1007/s00330-008-0880-6. Epub 2008 Feb 20. PMID 18286289
- [Background] Baek JH, Kim YS, Lee D, Huh JY, Lee JH. Benign predominantly solid thyroid nodules: prospective study of efficacy of sonographically guided radiofrequency ablation versus control condition. AJR Am J Roentgenol. 2010 Apr;194(4):1137-42. doi: 10.2214/AJR.09.3372. PMID 20308523
- [Background] Watt T, Barbesino G, Bjorner JB, Bonnema SJ, Bukvic B, Drummond R, Groenvold M, Hegedus L, Kantzer V, Lasch KE, Marcocci C, Mishra A, Netea-Maier R, Ekker M, Paunovic I, Quinn TJ, Rasmussen AK, Russell A, Sabaretnam M, Smit J, Torring O, Zivaljevic V, Feldt-Rasmussen U. Cross-cultural validity of the thyroid-specific quality-of-life patient-reported outcome measure, ThyPRO. Qual Life Res. 2015 Mar;24(3):769-80. doi: 10.1007/s11136-014-0798-1. Epub 2014 Sep 7. PMID 25194574
- [Background] Dobnig H, Amrein K. Monopolar Radiofrequency Ablation of Thyroid Nodules: A Prospective Austrian Single-Center Study. Thyroid. 2018 Apr;28(4):472-480. doi: 10.1089/thy.2017.0547. Epub 2018 Mar 20. PMID 29490593